CLINICAL TRIAL: NCT01588301
Title: Attitudes to Different Strategies Among Women Not Attending Cervical Cancer Screening: Further Invitation by Mail or Kit for Self-collected Vaginal Sample
Brief Title: Self-sampling and Human Papillomavirus (HPV)-Testing for Unscreened Women in Cervical Cancer Prevention
Acronym: APACHE-2
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: INCA08-KH / APACHE-2
Record Dates: First submitted 2012-03-12; First posted 2012-04-30 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-07

CONDITIONS: Cervical Cancer; Human Papillomavirus Infection
Keywords: Cervical Cancer Screening; Human Papillomavirus (HPV); Self-collected vaginal sample; Cervical Smear
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections | interventions — Receptor Protein-Tyrosine Kinases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 : Further invitation by mail (Experimental): Further invitation to attend for cervical cytology
  Interventions: Behavioral: Attending for cervical cytology
- Group 2 : Kit for Self-collected vaginal sample (Experimental): Kit for Self-collected vaginal sample sent at home and then test for Human Papillomavirus (HPV)
  Interventions: Behavioral: Kit for Self-collected vaginal sample
- Group 3: Control (No Intervention)

INTERVENTIONS:
Behavioral: Attending for cervical cytology — A further invitation to attend for cervical cytology are going to be sent by mail to women
  Arms: Group 1 : Further invitation by mail
Behavioral: Kit for Self-collected vaginal sample — Kit for self-collected vaginal sample are going to be directly sent at women's home
  Arms: Group 2 : Kit for Self-collected vaginal sample

SUMMARY:
Scientific Context:

High-risk types of human papillomavirus (HPV) are the causative agents for cervical cancer. Cervical cancer screening strategies rely on periodic Papanicolaou (Pap) testing. It's well-known that this test has significantly contributed to the reduction of mortality and morbidity due to cervical cancer. In France, it now seems that the screening strategy could be optimized. The two main ways are to reach the 7 million underscreened women (organized screening, self-sampling for HPV DNA testing) and to improve the screening test (HPV DNA testing, computer-assisted cytology). Self-collected vaginal samples (SCVS) for HPV DNA testing could be a relevant screening option: this technique appears reliable and it could allow to reach women who are never or seldom screened. The performance of the SCVS to detect cervical HPV infection has been assessed by the first part of the whole study: APACHE-1.

The goal of this study is to compare the attitudes of women not attending organized cervical cancer screening face to different strategies: further invitation to make a cervical smear or kit for self-collected vaginal sample sent at home.

Description of the project :

Nine months after a primary invitation to make a cervical smear, a random sample of 6000 women not attending organized cervical cancer screening will be randomly assigned to one of the following arms:

* Intervention arm 1:

Women will receive a further invitation to make a cervical smear

* Intervention arm 2:

Women will be directly sent the kit for self-collected vaginal sample at home. The women who will send the self-sample to the laboratory for analyse will receive their results at home as well as their general practitioner if the HPV DNA test is positive (infection by a high-risk HPV).

For them who will have a HPV DNA test positive, it will be necessary to complete the screening action with a cervical smear. That's why those women will receive an invitation to make a cervical smear if they won't do it during the 9 months following the first mail.

* Control arm: Those women will receive complete information about the study, the main results and the screening recommendations at the end of the study.

ELIGIBILITY:
Inclusion Criteria :

* Women from 30 to 65 years
* Living in Indre-et-Loire (french territorial division 37)

Exclusion Criteria :

* Women who attend organized cervical cancer screening or who answer to the invitation
* Cervical smear made in the three last years
* HPV linked cervical condition undergoing treatment
* Hysterectomy (including cervix)

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5998 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Comparison of women's attitude according to the arm: participation or not to a whole screening action | 9 months after the beginning of the study (sending of mails)
  Comparison of attitudes among women not attending organized cervical cancer according to the type of intervention or the lack of intervention: participation or not to a whole screening action.
  Are considered as whole screening action:
  * cervical smear
  * HPV DNA testing on self-collected vaginal sample negative (no infection by a high-risk HPV)
  * HPV DNA testing on self-collected vaginal sample positive (infection by a high-risk HPV) followed by a cervical smear

SECONDARY OUTCOMES:
Analysis in sub-groups | 9 months after the beginning of the study (sending of mails)
  Analysis in sub-groups in order to compare the efficacy of interventions according to :
  * The age
  * Health insurance system
  * Distribution map (urban area, peri-urban area, rural area)
Identification of the psychological determinants and mechanisms (checks and motivational factors) | 9 months after the beginning of the study (sending of mails)
  Identify the psychological determinants and mechanisms (checks and motivational factors) that can affect enrollment to the screening procedure for self-collection vaginal sample or cervical smear.
  Nine months after the beginning of the study, a questionnaire will be send to the 6000 women.

CONTACTS AND LOCATIONS:
Overall Officials: Ken HAGUENOER, Study Director — François Rabelais University, Public Health Laboratory, Tours, France